CLINICAL TRIAL: NCT03900468
Title: Medtronic Deep Brain Stimulation (DBS) Therapy for Epilepsy Post-Approval Study (EPAS)
Acronym: EPAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1677
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; Deep Brain Stimulation; DBS; EPAS
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Active Deep Brain Stimulation (DBS) (Experimental)
  Interventions: Device: Activa™ PC and Percept™ PC Neurostimulation Systems

INTERVENTIONS:
Device: Activa™ PC and Percept™ PC Neurostimulation Systems — Implanted DBS system consisting of a Neurostimulator, Leads, Extensions, and potential accessories including Burr Hole Devices, Clinician Tablet, Clinician Programmer Therapy Application Software, Clinician Programmer Communicator, Patient Programmer

SUMMARY:
The purpose of this post-approval study is to further evaluate the long-term safety and effectiveness of Medtronic DBS therapy for epilepsy on seizure reduction in newly implanted participants through 3 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Focal (partial) onset seizures (based on International League Against Epilepsy (ILAE) 2017 classification) that may or may not evolve to a bilateral tonic-clonic seizure (secondary generalization). The final determination shall be made by the Investigator based on a clinical description of the seizures and previous diagnostic testing that includes, at a minimum, video EEG (inpatient or ambulatory) that captured at least one ictal event
* Anticipated average of 6 or more focal (partial) onset seizures per month during CMM phase, with no more than 30 consecutive seizure-free days during the CMM phase
* Refractory to at least 3 antiepileptic drugs (AEDs) due to lack of effectiveness
* Age 18 or older at the time of enrollment
* Willing and able to complete the diary, with or without the assistance of a caregiver, in a reliable way as assessed by the clinical staff
* Able to use the Patient Programmer with or without the assistance of a caregiver
* Ability of the subject or legal representative to understand and provide signed consent for participating in the study
* Willing and available to attend visits as scheduled and to comply with the study protocol

Exclusion Criteria:

* Generalized onset epilepsy type (based on International League Against Epilepsy (ILAE) 2017 classification)
* Seizure frequency is too frequent that subject is unable to provide daily count in order to maintain a reliable seizure diary
* Any episode of convulsive status epilepticus within the 12 months prior to the Enrollment Visit
* Previous diagnosis of psychogenic/non-epileptic seizures within the 12 months prior to the Enrollment Visit
* Surgical candidate for and willing to undergo resective surgery
* Evidence of a neurological condition that is likely to progress (e.g., brain tumor, arteriovenous malformations or cavernous angiomas)
* Diagnosed with a progressive or degenerative neurological disorder affecting the brain
* Significant medical condition that may impact study participation in the opinion of the investigator
* Presence of any of the following within 1 year prior to the Enrollment Visit: psychiatric illness hospitalization, suicide attempt or symptoms of psychosis (hallucinations, delusions) unrelated to an ictal state, a post-ictal state or a medication
* Malignancy or history of malignancy within 1 year prior to the Enrollment Visit (excluding resected basal cell carcinomas)
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., cardiac pacemakers, spinal cord stimulator, RNS) or any metallic implants in the head (e.g., aneurysm clip, cochlear implant). In the case of an implanted vagus nerve stimulator (VNS), CMM study assessment collection may occur with the device implanted but may not begin until the VNS has been off for at least 30 days. The VNS generator must be explanted prior to or at the time of the DBS neurostimulator implant and the leads removed or trimmed and capped. In the case of a subject who had been previously implanted with a responsive neurostimulator (RNS) but had a full system explant, a subject cannot begin CMM study assessment collection until the RNS has been off for at least 30 days.
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. This includes administration of any antiplatelet or anticoagulant medication in the 7 days prior to surgery, chronic anticoagulant use, chronic aspirin use of greater than 325 mg/day, and any participant with a history of hemorrhagic stroke
* History of drug or alcohol abuse within the past year
* Condition or disease that is known to require repeat magnetic resonance imaging (MRIs)
* Currently participating, or plans to participate, in another investigational study unless written approval is provided by the Medtronic study team

Implant Criteria

* Experienced an average of 6 or more focal (partial) onset seizures per month during CMM phase, with no more than 30 consecutive seizure-free days (all seizure types)
* Completed a qualifying baseline diary. A qualifying baseline diary meets at least one the following criteria: 1) a study diary with at least 28 completed days; 2) a pre-existing diary with at least 70 completed days.
* Completed 3-month CMM visit
* No suicide attempt or other self-harm behaviors within past year (assessed by Columbia Suicide Severity Rating Scale (C-SSRS) at 3-month CMM Visit)
* For female subjects of child-bearing potential, has negative pregnancy test and if sexually active continues using reliable form of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2026-03-27 (Estimated)

PRIMARY OUTCOMES:
Percentage Reduction in Total Seizure Frequency | Pre-implant compared to 36 months post-implant
  The percentage of total seizure frequency reduction will be assessed using the participant seizure diaries to demonstrate DBS therapy effectiveness

SECONDARY OUTCOMES:
Percentage Reduction in Total Seizure Frequency | Pre-implant compared to 12 months post-implant
  The percentage of total seizure frequency reduction will be assessed using the participant seizure diaries to demonstrate DBS therapy effectiveness
Percentage Reduction in Total Disabling Seizure Frequency | Pre-implant compared to 12 months post-implant
  The percentage of total disabling seizure frequency reduction will be assessed using the participant seizure diaries to demonstrate DBS therapy effectiveness
Percentage Reduction in Temporal Lobe Originated Seizure Frequency | Pre-implant compared to 12 months post-implant
  The percentage of temporal lobe originated seizure frequency reduction will be assessed using the participant seizure diaries to demonstrate DBS therapy effectiveness
SUDEP Rate Characterization | Implant to 36 months post-implant
  To characterize the Sudden Unexplained Death in Epilepsy (SUDEP) rate. Any participant deaths will be reported in the study database and SUDEP will be evaluated and reported by the site. The Clinical Events Committee (CEC) will evaluate all deaths and make the final determination of SUDEP used for this objective.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of California San Francisco UCSF Medical Center, San Francisco, California
  - Stanford Hospital & Clinics, Stanford, California
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Health Neuroscience Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
- Fakultni nemocnice u sv. Anny v Brně/ Milan Brazdil, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No